CLINICAL TRIAL: NCT01103323
Title: A Randomized, Double-blind, Placebo-controlled Phase III Study of Regorafenib Plus BSC Versus Placebo Plus BSC in Patients With Metastatic Colorectal Cancer (CRC) Who Have Progressed After Standard Therapy
Brief Title: Patients With Metastatic Colorectal Cancer Treated With Regorafenib or Placebo After Failure of Standard Therapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14387; 2009-012787-14 (EudraCT Number)
Record Dates: First submitted 2010-04-08; First posted 2010-04-14 (Estimated); Results first posted 2012-11-19 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-05

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — regorafenib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regorafenib (Stivarga, BAY73-4506)+BSC (Experimental): Participants received Regorafenib 160 mg per oral once daily for 3 weeks on 1 week off of every 4 week cycle plus Best Supportive Care(BSC).
  Interventions: Drug: Regorafenib (Stivarga, BAY73-4506); Other: Best Supportive Care (BSC)
- Placebo+BSC (Placebo Comparator): Participants received matching placebo tablets per oral once daily for 3 weeks on 1 week off of every 4 week cycle plus Best Supportive Care (BSC).
  Interventions: Drug: Placebo; Other: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Regorafenib (Stivarga, BAY73-4506) — 160 mg per oral once daily for 3 weeks of every 4 week cycle (i.e., 3 weeks on, 1 week off)
  Arms: Regorafenib (Stivarga, BAY73-4506)+BSC
Drug: Placebo — matching placebo tablets for 3 weeks of every 4 week cycle (i.e., 3 weeks on, 1 week off)
  Arms: Placebo+BSC
Other: Best Supportive Care (BSC) — BSC includes any concomitant medications or treatments: antibiotics, analgesics, radiation therapy for pain control (limited to bone metastases), corticosteroids, transfusions, psychotherapy, growth factors, palliative surgery, or any other symptomatic therapy necessary to provide BSC, except other investigational anti-tumor agents or anti-neoplastic chemo/hormonal/immuno-therapy.

SUMMARY:
This is a randomized, double-blind, placebo-controlled multi-center phase III study to evaluate efficacy and safety of regorafenib in patients with metastatic colorectal cancer (CRC) who have progressed on/after all approved drugs for CRC

DETAILED DESCRIPTION:
All participants received Best Supportive Care. Acronyms used in Adverse events section: Gastrointestinal (GI), Genitourinary (GU), Not Otherwise Specified (NOS), Absolute Neutrophil Count (ANC), Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), Common Terminology Criteria for Adverse Events (CTCAE), International Normalized Ratio (INR), Central nervous system (CNS), Acute respiratory distress syndrome (ARDS), Cranial nerves (CN), Disseminated Intravascular Coagulation (DIC), Cardiac troponin T (cTnT).

Abbreviation used in Results section: Data Monitoring Committee (DMC). Adverse event collection will be covered in Adverse events section.

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological documentation of adenocarcinoma of the colon or rectum
* Progression during or within 3 months following the last administration of approved standard therapies. Patients treated with oxaliplatin in an adjuvant setting should have progressed during or within 6 months of completion of adjuvant therapy
* Patients with measurable or non measurable disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of </= 1
* Life expectancy of at least 3 months
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Unstable/uncontrolled cardiac disease
* History of arterial or venous thrombotic or embolic events
* Symptomatic metastatic brain or meningeal tumors
* Patients with evidence or history of bleeding diathesis
* Interstitial lung disease - Persistent proteinuria >/= grade 3
* Unresolved toxicity > grade 1 attributed to any prior therapy/procedure excluding alopecia and oxaliplatin induced neurotoxicity </= Grade 2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 760 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (155):
- United States (25):
  - Beverly Hills, California
  - Los Angeles, California
  - Mission Hills, California
  - Orange, California
  - Redlands, California
  - Santa Maria, California
  - Aventura, Florida
  - Jacksonville, Florida
  - Peoria, Illinois
  - Cedar Rapids, Iowa
  - New Orleans, Louisiana
  - Ann Arbor, Michigan
  - Rochester, Minnesota
  - Saint Cloud, Minnesota
  - Jefferson City, Missouri
  - Neptune City, New Jersey
  - New York, New York
  - Fargo, North Dakota
  - Toledo, Ohio
  - Scranton, Pennsylvania
  - Charleston, South Carolina
  - Sumter, South Carolina
  - Dallas, Texas
  - Salt Lake City, Utah
  - Green Bay, Wisconsin
- Argentina (4):
  - Buenos Aires, Ciudad Auton. de Buenos Aires
  - Rosario, Santa Fe Province
  - San Miguel de Tucumán, Tucumán Province
  - Capital Federal-Buenos Aires
- Australia (6):
  - Concord, New South Wales
  - St Leonards, New South Wales
  - Woolloogabba, Queensland
  - Woodville South, South Australia
  - Footscray, Victoria
  - Parkville, Victoria
- Belgium (4):
  - Bruxelles - Brussel
  - Edegem
  - Leuven
  - Roeselare
- Brazil (4):
  - Fortaleza, Ceará
  - Salvador, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Ijuí, Rio Grande do Sul
- Canada (9):
  - Vancouver, British Columbia
  - Winnipeg, Manitoba
  - Moncton, New Brunswick
  - London, Ontario
  - Mississauga, Ontario
  - Oshawa, Ontario
  - Toronto, Ontario
  - Montreal, Quebec
  - Québec, Quebec
- China (11):
  - Guangzhou, Guangdong
  - Nanjing, Jiangsu
  - Qingdao, Shandong
  - Beijing
  - Changchun
  - Chongqing
  - Fuzhou
  - Hanghzou
  - Ha’erbin
  - Shanghai
  - Tianjin
- Czechia (4):
  - Brno
  - Hradec Králové
  - Olomouc
  - Prague
- France (10):
  - Lille, Lille Cedex
  - Avignon
  - Le Mans
  - Lille
  - Marseille
  - Montpellier
  - Paris
  - Reims
  - Rennes
  - Strasbourg
- Germany (16):
  - Freiburg im Breisgau, Baden-Wurttemberg
  - Karlsruhe, Baden-Wurttemberg
  - Mannheim, Baden-Wurttemberg
  - Stuttgart, Baden-Wurttemberg
  - München, Bavaria
  - Hanover, Lower Saxony
  - Oldenburg, Lower Saxony
  - Cologne, North Rhine-Westphalia
  - Essen, North Rhine-Westphalia
  - Leverkusen, North Rhine-Westphalia
  - Porta Westfalica, North Rhine-Westphalia
  - Trier, Rhineland-Palatinate
  - Dresden, Saxony
  - Halle, Saxony-Anhalt
  - Magdeburg, Saxony-Anhalt
  - Berlin, State of Berlin
- Hungary (4):
  - Budapest
  - Debrecen
  - Nyíregyháza
  - Szeged
- Israel (10):
  - Zrifin, Israel
  - Ashkelon
  - Beersheba
  - Haifa
  - Holon
  - Jerusalem
  - Petah Tikva
  - Rehovot
  - Tel Aviv
  - Tel Litwinsky
- Italy (8):
  - Brescia
  - Genova
  - Milan
  - Modena
  - Napoli
  - Pisa
  - Reggio Emilia
  - Roma
- Japan (20):
  - Nagoya, Aichi-ken
  - Chiba, Chiba
  - Kashiwa, Chiba
  - Matsuyama, Ehime
  - Fukuoka, Fukuoka
  - Sapporo, Hokkaido
  - Kochi, Kochi
  - Kumamoto, Kumamoto
  - Osaka, Osaka
  - Sayama, Osaka
  - Takatsuki, Osaka
  - Hidaka, Saitama
  - Kita-Adachigun, Saitama
  - Sunto, Shizuoka
  - Shimotsuke, Tochigi
  - Utsunomiya, Tochigi
  - Bunkyo-ku, Tokyo
  - Chuo-ku, Tokyo
  - Koto-ku, Tokyo
  - Mitaka, Tokyo
- Netherlands (4):
  - Amsterdam
  - Hoofddorp
  - Leeuwarden
  - Leiden
- Portugal (4):
  - Aveiro, Aveiro District
  - Porto, Porto District
  - Coimbra
  - Lisbon
- Spain (6):
  - Barcelona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Sabadell, Barcelona
  - Madrid, Madrid
  - Málaga, Málaga
  - Seville, Sevilla
- Switzerland (2):
  - Geneva, Canton of Geneva
  - Chur, Kanton Graubünden
- Turkey (Türkiye) (4):
  - Ankara
  - Instanbul
  - Istanbul
  - Izmir

REFERENCES:
- [Result] Grothey A, Van Cutsem E, Sobrero A, Siena S, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Tabernero J, Yoshino T, Lenz HJ, Goldberg RM, Sargent DJ, Cihon F, Cupit L, Wagner A, Laurent D; CORRECT Study Group. Regorafenib monotherapy for previously treated metastatic colorectal cancer (CORRECT): an international, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2013 Jan 26;381(9863):303-12. doi: 10.1016/S0140-6736(12)61900-X. Epub 2012 Nov 22. PMID 23177514
- [Result] Mross K, Frost A, Steinbild S, Hedbom S, Buchert M, Fasol U, Unger C, Kratzschmar J, Heinig R, Boix O, Christensen O. A phase I dose-escalation study of regorafenib (BAY 73-4506), an inhibitor of oncogenic, angiogenic, and stromal kinases, in patients with advanced solid tumors. Clin Cancer Res. 2012 May 1;18(9):2658-67. doi: 10.1158/1078-0432.CCR-11-1900. Epub 2012 Mar 15. PMID 22421192
- [Derived] Cervantes A, Tabernero J, Garcia-Carbonero R, Sastre J, Feliu J, Carmen Guillen-Ponce, Paredes BG, Carral A, Munoz J. Regorafenib in patients with metastatic colorectal cancer in Spain: from clinical trials to real-world evidence. Future Oncol. 2024;20(20):1401-1413. doi: 10.1080/14796694.2024.2340422. Epub 2024 Jun 11. PMID 38861286
- [Derived] Tabernero J, Lenz HJ, Siena S, Sobrero A, Falcone A, Ychou M, Humblet Y, Bouche O, Mineur L, Barone C, Adenis A, Yoshino T, Goldberg RM, Sargent DJ, Wagner A, Laurent D, Teufel M, Jeffers M, Grothey A, Van Cutsem E. Analysis of circulating DNA and protein biomarkers to predict the clinical activity of regorafenib and assess prognosis in patients with metastatic colorectal cancer: a retrospective, exploratory analysis of the CORRECT trial. Lancet Oncol. 2015 Aug;16(8):937-48. doi: 10.1016/S1470-2045(15)00138-2. Epub 2015 Jul 13. PMID 26184520
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Groups:
- Regorafenib (Stivarga, BAY73-4506)+BSC: Participants received Regorafenib 160 mg per oral once daily for 3 weeks on 1 week off of every 4 week cycle plus best supportive care (BSC).
- Placebo+BSC: Participants received matching placebo tablets per oral once daily for 3 weeks on 1 week off of every 4 week cycle plus best supportive care (BSC). Period 1 is placebo and placebo-regorafenib with placebo period only before unblinding. Period 2 is placebo-regorafenib with regorafenib period only.
Period: Without/Before Drug Switch
Arm/Group | Regorafenib (Stivarga, BAY73-4506)+BSC | Placebo+BSC
Started | 505 | 255
Participants Received Treatment | 500 | 253
Completed | 429 | 237
Not Completed | 76 | 18
Not completed — Adverse Event | 50 | 7
Not completed — Withdrawal by Subject | 17 | 5
Not completed — Protocol Violation | 2 | 0
Not completed — Physician Decision | 2 | 0
Not completed — did not receive study treatment | 5 | 2
Not completed — Switch to Regorafenib | 0 | 4
Period: Switched From Placebo to Regorafenib
Arm/Group | Regorafenib (Stivarga, BAY73-4506)+BSC | Placebo+BSC
Started | 0 | 4 (Participants in the placebo+BSC group switched to Regorafenib treatment after unblinding.)
Completed | 0 | 3
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Regorafenib (Stivarga, BAY73-4506)+BSC | Placebo+BSC | Total
Number analyzed (Participants) | 505 | 255 | 760
Age, Continuous [Mean (Full Range); unit: Years] — The age of the patient in years at enrollment in the study.
  Years | 60.7 [22 to 82] | 60.1 [25 to 85] | 60.5 [22 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 194 | 102 | 296
  Male | 311 | 153 | 464
Eastern Cooperative Oncology Group (ECOG) performance status (PS) before treatment [Number; unit: Participants] — ECOG PS is a scale that measures how cancer affects the daily life of a patient on an ordinal scale from grade 0 (best) to grade 5 (worst). 0=Fully active without restriction; 1= Restricted in physically strenuous activity; 2= Ambulatory, capable of all selfcare; 3= Capable of limited selfcare; 4= Completely disabled; 5= Dead
  Participants
    0 | 265 | 146 | 411
    1 | 240 | 109 | 349
KRAS mutation [Number; unit: Participants] — KRAS - Kirsten rat sarcoma viral oncogene homolog (protein), member of the RAS family of GTPases (guanosine triphosphate hydrolases)
  Participants
    No | 205 | 94 | 299
    Yes | 273 | 157 | 430
    Unknown | 27 | 4 | 31

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) was defined as the time (days) from randomization to death due to any cause. Patients alive at the time of analysis were censored at the last date known to be alive. If a patient was lost to follow-up and there was no contact after randomization, this patient was censored at Day 1.
Time Frame: From randomization of the first subject until the database cut-off approximately 14 months later (19May2010 - 21Jul2011) used for 2nd planned formal interim analysis (IA).
Population: Intent to treat (ITT)
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)+BSC | Placebo+BSC
Number analyzed (Participants) | 505 | 255
Days | 196 [178 to 222] | 151 [134 to 177]
Statistical Analysis 1: Comparison: Regorafenib (Stivarga, BAY73-4506)+BSC vs Placebo+BSC; Sample size based on primary efficacy endpoint of OS. The study was designed to have 90% power to detect 33.3% increase in median OS (i.e. hazard ratio of 0.75, Regorafenib / Placebo). Assuming 1-sided overall alpha of 0.025, randomization ratio of 2:1 for Regorafenib and Placebo, and 2 formal interim analyses of OS using an O'Brien-Fleming-type error spending function, a total of 582 death events were required for primary completion. Results based on 2nd planned formal IA with 432 total events; Test type: Superiority or Other; p = 0.005178, Log Rank — According to protocol specified O'Brien-Fleming type alpha spending function and 432 death events at 2nd IA, the pre-specified alpha (false positive rate) for this analysis was 0.009279 (1-sided); Hazard Ratio (HR) = 0.774, 95% CI [0.636 to 0.942] — Two treatment groups compared using a stratified log-rank test, stratified by same stratification factors as randomization. Hazard ratio (Regorafenib / Placebo) and its 95% confidence interval calculated using Cox model, stratified by same factors

2. Secondary Outcome: Progression-free Survival (Based on Investigator's Assessment)
Description: Progression-free survival was defined as the time (days) from date of randomization to date of first observed disease progression (radiological or clinical) or death due to any cause, if death occurred before progression was documented.
Time Frame: From randomization of the first subject until the database cut-off approximately 14 months later (19May2010 - 21Jul2011) used for 2nd planned formal interim analysis. Tumor assessed at 8 week intervals.
Population: ITT
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Regorafenib (Stivarga, BAY73-4506)+BSC | Placebo+BSC
Number analyzed (Participants) | 505 | 255
Days | 59 [57 to 65] | 52 [51 to 53]
Statistical Analysis 1: Comparison: Regorafenib (Stivarga, BAY73-4506)+BSC vs Placebo+BSC; Two treatment groups compared using a stratified log-rank test, stratified by same stratification factors as randomization. Hazard ratio (Regorafenib / Placebo) and its 95% confidence interval calculated using Cox model, stratified by same factors; Test type: Superiority or Other; p < 0.000001, Log Rank — Comparison based on pre-specified alpha level of 0.025 (1-sided); Hazard Ratio (HR) = 0.494, 95% CI [0.419 to 0.582] — Hazard ratio (Regorafenib / Placebo)

3. Secondary Outcome: Objective Tumor Response
Description: The objective tumor response was defined as the percentage of patients with complete response (CR, tumor disappears) or partial response (PR, sum of lesion sizes decreased at least 30% from baseline) as best overall response. A best overall response was defined for all patients, using the Response Evaluation Criteria in Solid Tumors (RECIST) criteria, version 1.1. Patients whose best overall response was not CR or PR, and any patients with no post-baseline assessments were considered nonresponders for the analysis.
Time Frame: as for outcome 2
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506)+BSC | Placebo+BSC
Number analyzed (Participants) | 505 | 255
Percentage of participants | 1.0 | 0.4
Statistical Analysis 1: Comparison: Regorafenib (Stivarga, BAY73-4506)+BSC vs Placebo+BSC; Two treatment groups compared using Cochran-Mantel-Haenszel (CMH) test adjusting for same stratification factors as at randomization; Test type: Superiority or Other; p = 0.188432, Cochran-Mantel-Haenszel — Comparison based on pre-specified alpha level of 0.025 (1-sided); Difference = -0.60, 95% CI [-1.74 to 0.53] — Difference = Placebo - Regorafenib 160 mg

4. Secondary Outcome: Disease Control
Description: Disease control was defined as the percentage of patients whose best response was not PD [sum of lesion sizes increased at least 20% from smallest sum on study or new lesions] (ie, CR [tumor disappears], PR [sum of lesion sizes decreased at least 30% from baseline] or SD (stable disease)). SD included if at least 6 weeks after randomization.
Time Frame: as for outcome 2
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506)+BSC | Placebo+BSC
Number analyzed (Participants) | 505 | 255
Percentage of participants | 41.0 | 14.9
Statistical Analysis 1: Comparison: Regorafenib (Stivarga, BAY73-4506)+BSC vs Placebo+BSC; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.000001, Cochran-Mantel-Haenszel — Comparison based on pre-specified alpha level of 0.025 (1-sided); Difference = -25.94, 95% CI [-32.06 to -19.82] — Difference = Placebo - Regorafenib 160 mg

5. Secondary Outcome: Tumor Response
Description: A tumor response (best overall response) was defined for all patients, using the RECIST criteria, version 1.1. Categories: complete response (CR, tumor disappears), partial response (PR, sum of lesion sizes decreased at least 30% from baseline), stable disease (SD, steady state of disease), progressive disease (PD, sum of lesion sizes increased at least 20% from smallest sum on study or new lesions). Clinical PD considered when radiographic imaging not possible.
Time Frame: as for outcome 2
Population: ITT
Measure: Number; unit: Percentage of participants
Arm/Group | Regorafenib (Stivarga, BAY73-4506)+BSC | Placebo+BSC
Number analyzed (Participants) | 505 | 255
Percentage of participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 1.0 | 0.4
  Stable Disease (SD) | 42.8 | 14.5
  Progressive Disease (PD) | 49.5 | 80.0
  Non CR/Non PD | 0.8 | 0.4
  Not applicable | 0.2 | 0
  Not assessed | 5.7 | 4.7

ADVERSE EVENTS:
Time Frame: AE was collected up to 30 days after end of study treatment (per protocol) over a period of approximately 3.7 years.
Description: Disseminated Intravascular Coagulation (DIC), International Normalized Ratio (INR), Cardiac Troponin T (cTnT), Gastroihntestina (GI), Not Otherwise Specified (NOS), Aspartate Aminotransferase (AST), Genitourinary (GU), Alanine Aminotransferase (ALT), Acute Respiratory Distress Syndrome (ARDS), Absolute Neutrophil Count (ANC)
Groups:
- Regorafenib (BAY73-4506)+BSC: Participants received Regorafenib 160 mg per oral once daily for 3 weeks on 1 week off of every 4 week cycle plus best supportive care (BSC).
- Placebo+BSC: Participants received matching placebo tablets per oral once daily for 3 weeks on 1 week off of every 4 week cycle plus best supportive care (BSC). It is for placebo period only before unblinding.
- Placebo - Regorafenib After Unblinding: Participants in the placebo+BSC group switched to treatment with Regorafenib after unblinding. It is for Regorafenib treatment period only
Arm/Group | Regorafenib (BAY73-4506)+BSC | Placebo+BSC | Placebo - Regorafenib After Unblinding
Serious Adverse Events (participants affected / at risk) | 232/500 | 103/253 | 2/4
Other Adverse Events (participants affected / at risk) | 489/500 | 229/253 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (BAY73-4506)+BSC (N=500) | Placebo+BSC (N=253) | Placebo - Regorafenib After Unblinding (N=4)
DIC (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Edema: Limb (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 0 (0)
Edema: Trunk/Genital (Blood and lymphatic system disorders) | 0 (0) | 2 (4) | 0 (0)
Edema: Viscera (Blood and lymphatic system disorders) | 0 (0) | 1 (3) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 4 (8) | 2 (2) | 0 (0)
INR (Blood and lymphatic system disorders) | 2 (5) | 0 (0) | 0 (0)
Neutrophils (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrhythmia - Other (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac ischemia/infarction (Cardiac disorders) | 6 (6) | 1 (2) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (3) | 0 (0) | 0 (0)
Supraventricular arrhythmia, Atrial fibrillation (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
cTnT (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 1 (1) | 0 (0)
Ocular - Other (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Anorexia (Gastrointestinal disorders) | 5 (8) | 2 (2) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 2 (2) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 8 (9) | 0 (0) | 0 (0)
Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fistula, GI, Abdomen NOS (Gastrointestinal disorders) | 1 (2) | 1 (1) | 0 (0)
Fistula, GI, Anus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Fistula, GI, Small bowel NOS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
GI - Other (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 2 (3) | 3 (3) | 0 (0)
Mucositis (functional/symptomatic), Small bowel (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Necrosis, GI, Peritoneal cavity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Obstruction, GI, Colon (Gastrointestinal disorders) | 9 (11) | 6 (8) | 0 (0)
Obstruction, GI, Ileum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Obstruction, GI, Small bowel NOS (Gastrointestinal disorders) | 4 (5) | 7 (9) | 0 (0)
Obstruction, GI, Stomach (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Perforation, GI, Colon (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stricture, GI, Biliary tree (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Ulcer, GI, Duodenum (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Constitutional symptoms - Other (General disorders) | 34 (49) | 23 (39) | 0 (0)
Death not associated with CTCAE term, Disease progression NOS (General disorders) | 16 (17) | 6 (6) | 1 (1)
Death not associated with CTCAE term, Multi-Organ Failure (General disorders) | 4 (4) | 1 (1) | 0 (0)
Death not associated with CTCAE term, Sudden death (General disorders) | 2 (2) | 2 (2) | 0 (0)
Fatigue (General disorders) | 5 (6) | 5 (5) | 0 (0)
Fever (General disorders) | 17 (21) | 2 (2) | 0 (0)
Pain, Abdomen NOS (General disorders) | 13 (21) | 2 (2) | 0 (0)
Pain, Back (General disorders) | 4 (6) | 4 (5) | 0 (0)
Pain, Buttock (General disorders) | 2 (4) | 0 (0) | 0 (0)
Pain, Cardiac/Heart (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain, Chest wall (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain, Chest/Thorax NOS (General disorders) | 4 (4) | 1 (1) | 0 (0)
Pain, Extremity - limb (General disorders) | 2 (6) | 0 (0) | 0 (0)
Pain, Head/Headache (General disorders) | 2 (2) | 1 (1) | 0 (0)
Pain, Joint (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain, Liver (General disorders) | 1 (2) | 0 (0) | 0 (0)
Pain, Neuralgia/Peripheral nerve (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pain, Pain NOS (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pain, Tumor pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Syndromes - Other (General disorders) | 1 (1) | 0 (0) | 0 (0)
Tumor flare (General disorders) | 1 (2) | 0 (0) | 0 (0)
Weight loss (General disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Hepatobiliary - Other (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0)
Liver dysfunction (Hepatobiliary disorders) | 17 (28) | 5 (11) | 0 (0)
Allergic reaction (Immune system disorders) | 2 (4) | 0 (0) | 0 (0)
Infection (documented clinically), Abdomen NOS (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Infection (documented clinically), Anal/perianal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (documented clinically), Appendix (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (documented clinically), Bladder (urinary) (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Infection (documented clinically), Blood (Infections and infestations) | 3 (5) | 2 (2) | 0 (0)
Infection (documented clinically), Bronchus (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Infection (documented clinically), Catheter-related (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Infection (documented clinically), Kidney (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection (documented clinically), Lung (Pneumonia) (Infections and infestations) | 9 (11) | 3 (4) | 0 (0)
Infection (documented clinically), Skin (Cellulitis) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (documented clinically), Soft tissue NOS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection (documented clinically), Urinary tract NOS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infection (documented clinically), Wound (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection - Other (Infections and infestations) | 5 (6) | 1 (2) | 0 (0)
Infection with normal ANC, Blood (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC, Catheter-related (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC, Colon (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC, Gallbladder (Cholecystitis) (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC, Kidney (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC, Lung (Pneumonia) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection with normal ANC, Soft tissue NOS (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Infection with unknown ANC, Kidney (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with unknown ANC, Lung (Pneumonia) (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
AST (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 8 (11) | 3 (3) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Fracture (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (3) | 0 (0)
Gait/Walking (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Muscle weakness left-sided (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle weakness, Extremity - lower (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Muscle weakness, Whole body/generalized (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal - Other (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Secondary malignancy (possibly related to cancer treatment) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 (0) | 0 (0)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
CNS ischemia (Nervous system disorders) | 1 (2) | 2 (2) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Mood Alteration, Anxiety (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0)
Neurology - Other (Nervous system disorders) | 3 (4) | 2 (2) | 0 (0)
Neuropathy: Cranial, CN III Pupil, upper eyelid, extra ocular mov (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Neuropathy: motor (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Speech impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Fainting) (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Cystitis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Fistula, GU, Bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Obstruction, GU, Ureter (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0)
Renal - Other (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 5 (6) | 3 (5) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 2 (2) | 0 (0)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 12 (18) | 4 (4) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 4 (4) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Pulmonary - Other (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3) | 0 (0)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 1 (3) | 0 (0) | 0 (0)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 4 (7) | 1 (1) | 0 (0)
Wound complication, non-infectious (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Hematoma (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage - Other (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage pulmonary, Bronchus (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Hemorrhage pulmonary, Mediastinum (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI, Abdomen NOS (Vascular disorders) | 2 (4) | 0 (0) | 0 (0)
Hemorrhage, GI, Anus (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Hemorrhage, GI, Lower GI NOS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI, Rectum (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI, Stoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI, Upper GI NOS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GI, Varices (esophageal) (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hemorrhage, GI, Varices (rectal) (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Hemorrhage, GU, Vagina (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Thrombosis/Embolism (vascular access) (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombosis/Thrombus/Embolism (Vascular disorders) | 6 (6) | 3 (5) | 0 (0)
Vascular - Other (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Regorafenib (BAY73-4506)+BSC (N=500) | Placebo+BSC (N=253) | Placebo - Regorafenib After Unblinding (N=4)
Edema: Limb (Blood and lymphatic system disorders) | 49 (57) | 16 (19) | 0 (0)
Hemoglobin (Blood and lymphatic system disorders) | 76 (142) | 29 (46) | 0 (0)
Platelets (Blood and lymphatic system disorders) | 79 (136) | 6 (9) | 1 (2)
Hypertension (Cardiac disorders) | 155 (213) | 21 (23) | 1 (1)
Hypothyroidism (Endocrine disorders) | 27 (29) | 1 (1) | 1 (1)
Ocular - Other (Eye disorders) | 5 (5) | 0 (0) | 1 (1)
Anorexia (Gastrointestinal disorders) | 239 (388) | 73 (96) | 0 (0)
Ascites (Gastrointestinal disorders) | 23 (24) | 6 (8) | 1 (1)
Constipation (Gastrointestinal disorders) | 119 (147) | 48 (58) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 218 (514) | 44 (57) | 2 (2)
Fistula, GI, Colon/Cecum/Appendix (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Mucositis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 145 (267) | 12 (12) | 0 (0)
Nausea (Gastrointestinal disorders) | 115 (162) | 55 (67) | 1 (1)
Taste alteration (Gastrointestinal disorders) | 39 (44) | 6 (6) | 0 (0)
Vomiting (Gastrointestinal disorders) | 85 (144) | 41 (50) | 1 (3)
Constitutional symptoms - Other (General disorders) | 30 (33) | 17 (19) | 0 (0)
Fatigue (General disorders) | 318 (612) | 115 (168) | 0 (0)
Fever (General disorders) | 136 (189) | 40 (48) | 2 (3)
Flu-like syndrome (General disorders) | 27 (30) | 6 (8) | 1 (1)
Insomnia (General disorders) | 39 (43) | 14 (15) | 0 (0)
Pain, Abdomen NOS (General disorders) | 121 (239) | 47 (53) | 0 (0)
Pain, Back (General disorders) | 79 (114) | 25 (27) | 0 (0)
Pain, Buttock (General disorders) | 4 (5) | 0 (0) | 1 (1)
Pain, Chest/Thorax NOS (General disorders) | 26 (29) | 12 (14) | 0 (0)
Pain, Extremity - limb (General disorders) | 51 (83) | 14 (19) | 0 (0)
Pain, Head/Headache (General disorders) | 50 (65) | 18 (23) | 0 (0)
Pain, Joint (General disorders) | 32 (34) | 13 (14) | 0 (0)
Pain, Muscle (General disorders) | 50 (64) | 14 (16) | 0 (0)
Pain, Throat/Pharynx/Larynx (General disorders) | 9 (12) | 1 (1) | 1 (1)
Weight loss (General disorders) | 167 (240) | 30 (34) | 2 (7)
Hepatobiliary - Other (Hepatobiliary disorders) | 8 (9) | 4 (4) | 1 (3)
ALT (Metabolism and nutrition disorders) | 28 (53) | 7 (8) | 0 (0)
AST (Metabolism and nutrition disorders) | 37 (72) | 12 (13) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 35 (49) | 8 (12) | 0 (0)
Bilirubin (Hyperbilirubinemia) (Metabolism and nutrition disorders) | 97 (160) | 22 (37) | 1 (3)
Creatinine (Metabolism and nutrition disorders) | 15 (19) | 7 (8) | 1 (2)
GFR (Metabolism and nutrition disorders) | 4 (9) | 1 (2) | 1 (1)
Hyperuricemia (Metabolism and nutrition disorders) | 12 (13) | 1 (1) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 34 (57) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 50 (84) | 6 (7) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 32 (43) | 6 (10) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 32 (62) | 2 (3) | 1 (2)
Lipase (Metabolism and nutrition disorders) | 32 (74) | 3 (4) | 0 (0)
Metabolic/Lab - Other (Metabolism and nutrition disorders) | 42 (69) | 8 (15) | 0 (0)
Proteinuria (Metabolism and nutrition disorders) | 40 (109) | 6 (11) | 0 (0)
Dizziness (Nervous system disorders) | 28 (31) | 13 (13) | 0 (0)
Neuropathy: sensory (Nervous system disorders) | 51 (68) | 25 (27) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 56 (77) | 28 (32) | 1 (1)
Dyspnea (Shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 89 (110) | 34 (46) | 0 (0)
Voice changes (Respiratory, thoracic and mediastinal disorders) | 160 (211) | 16 (17) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 39 (43) | 4 (4) | 0 (0)
Cheilitis (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0) | 1 (3)
Dermatology - Other (Skin and subcutaneous tissue disorders) | 30 (45) | 7 (10) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 50 (59) | 10 (11) | 0 (0)
Hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 235 (720) | 19 (21) | 1 (3)
Pruritus (Skin and subcutaneous tissue disorders) | 29 (39) | 11 (11) | 0 (0)
Rash/Desquamation (Skin and subcutaneous tissue disorders) | 145 (211) | 13 (17) | 1 (2)
Hemorrhage pulmonary, Nose (Vascular disorders) | 45 (55) | 6 (6) | 0 (0)

LIMITATIONS AND CAVEATS:
At 2nd IA, pre-specified O'Brien-Fleming-type efficacy boundary was crossed. DMC concluded OS result positive and after positive risk benefit assessment, recommended unblinding of study. OS from 2nd IA are the final formal and definitive results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The agreed point of publication is 12-18 months after database lock at the earliest. Bayer will have 30-45 days to review publications, and may request an additional publication delay of up to 60 days to allow for filing a Patent Application (if applicable). No publication of single center data should be done prior of publication if multi-center data.